

#### PHARMACOKINETIC DATA ANALYSIS PLAN

A randomized, open label, two-part, parallel-group, phase I study to evaluate the pharmacokinetics of Piperaquine oral dispersible Granules Formulation compared to Piperaquine hard Tablets administered as a single dose in fasting condition (Part 1) and of Piperaquine oral dispersible Granules Formulation administered as single dose in various fed states (Part 2) in healthy adult participants

PharmaKinetic Study Number: PHK2020-174

**Sponsor Study Number:** MMV\_SMC\_22\_01

**Sponsor:** Medicines for Malaria Venture (MMV)

ICC – Block G, 3rd floor 20, Route de Pré-Bois

PO Box 1826 1215 Geneva 15 Switzerland

**Date of Analysis Plan:** 02<sup>nd</sup> October 2023

**Version Number:** Version 2.0

# **Approval Signatures**

This PK analysis plan has been approved by.

# On behalf of Sponsor,



anne Claire Marrast

U

Signer Name: Anne Claire Marrast Signing Reason: I approve this document Signing Time: 03-Oct-23 | 1:52 PM BST -EE083864215049D7B3D27D3273F6C88A DocuSigned by:

Denis Gossen

Signer Name: Denis Gossen Signing Reason: I approve this document Signing Time: 02-Oct-23 | 5:35 PM BST -AC827ABF3B454D26A93B7F2C91B125E9

# On behalf of PharmaKinetic,

DocuSigned by:

Rachael White



Signer Name: Rachael White

Signing Reason: I approve this document Signing Time: 02-Oct-23 | 10:37 AM BST -2BDFAD0FF6B34023A90E30CE7A0ABDD0

# 1 Document Version History

| Version Number | Reason for Update | Updated By: | Date |
|---|---|---|---|
| Version 1.0 | First version issue | Rachael White | 8 <sup>th</sup> August 2023 |
| Version 2.0 | Version updated to include AUC(0-24) as a required PK parameter | Rachael White | 2 <sup>nd</sup> October 2023 |

# **Table of Contents**

| 1 | Docume | ent Version History | 2 |
|---|---|---|---|
| 2 | Table of | Contents | 3 |
| 3 | Study D | esign | 4 |
| | 3.1 | Outline Design and Pharmacokinetic Objectives | 4 |
| | 3.1.1 | Pharmacokinetic Objectives | 4 |
| | 3.1.2 | Pharmacokinetic Endpoints | 5 |
| 4 | Populati | ons for Analysis | 5 |
| | 4.1 | Pharmacokinetic Population | 5 |
| 5 | Pharmac | cokinetic Data Analysis | 5 |
| | 5.1 | Pharmacokinetic Parameter Estimation | 5 |
| | 5.1.1 | Imputation of Non-Numerical or Negative Values | 5 |
| | 5.1.2 | Rules for Pharmacokinetic Parameter Estimation using WinNonlin | 6 |
| | 5.1.3 | Data Quality | 6 |
| | 5.1.4 | Definition of Pharmacokinetic Parameters | 6 |
| | 5.2 | Statistical Analysis | 8 |
| | 5.3 | Interim Analysis | 8 |

# 3 Study Design

# 3.1 Outline Design and Pharmacokinetic Objectives

This is a randomized, open label, parallel-design study to evaluate the PK profile and relative bioavailability of single dose of a PQP oral granule formulation dispersed in water (test) as compared to the PQP hard tablet formulation (reference) in fasting conditions (Part 1) and to assess the BA/FE of the PQP dispersible granules formulation when administered with different food restrictions (Part 2) among African participants residing in Tanzania, in Bagamoyo Town and surrounding areas. A total of sixty (60) healthy adult participants (male and female) will be enrolled in Part 1 and Part 2.

Part 1: PQP tablet / dispersible granule administered in fasting condition of at least 10 hours

- Group 1: PQP hard tablet, 320 mg (N=12)
- Group 2: PQP dispersible granule, 320 mg (N=12)

#### Transition to Part 2:

• To minimize the risk to healthy participants, a decision on transitioning from Part 1 to Part 2, will be taken by the Safety Review Committee (SRC), based on the safety and preliminary PK interim report of the granule formulation, compared to the PQP hard tablet, with safety data obtained up to Day 15 and PK data obtained up to Day 8. If necessary, doses may be readjusted for the Part 2 in order to assess the food effect, to ensure that the predicted exposure of PQP from the granule formulation in the fed state doesn't exceed the exposure achieved in adults administered a dose of 960 mg PQP in a tablet of Eurartesim® in fasted conditions. Note, the observed food effect when film-coated tablets (Eurartesim®) are administered with a high fat/high calorie meal is a 3-fold increase in exposure.

Part 2: PQP dispersible granule administered in fed conditions (planned as 320 mg)

- Group 3: High-fat meal (N=12)
- Group 4: Low-fat meal representative of African diet (N=12)
- Group 5: Whole milk 250 ml (N=12)

# 3.1.1 Pharmacokinetic Objectives

# Primary:

• To determine the relative bioavailability of a single oral dose of PQP dispersible granule formulation (Test) as compared to POP hard tablet formulation (Reference) in the fasted state.

# Secondary:

- To assess the effect of different types of meal composition on the PK of single doses of PQP dispersible granule formulation in healthy adult participants.
- To further evaluate the PK of a single oral dose of PQP granule formulation in the fasted state and different fed states in healthy adult participants.

# 3.1.2 Pharmacokinetic Endpoints

# Primary:

• Relative bioavailability (F<sub>rel</sub>) using the ratio of the geometric means for the dispersible granule (test) over the hard tablet (reference) in fasted state for area under the plasma concentration-time curve from time zero to 72 hours (AUC<sub>0-72h</sub>), area under the plasma concentration-time curve from time zero to last detectable plasma concentration (AUC<sub>0-1</sub>), area under the plasma concentration-time curve from time zero to 168 hours (AUC<sub>0-168h</sub>), area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC<sub>0-∞</sub>), and Maximum plasma concentration (C<sub>max</sub>).

# Secondary

- The F<sub>rel</sub> using the ratio of the geometric means for the dispersible granules formulation between fed [high-fat meal, low-fat African meal, and milk] over the dispersible granule formulation fasted [reference] for AUC<sub>0-72h</sub>, AUC<sub>0-t</sub>, AUC<sub>0-168h</sub>, AUC<sub>0-∞</sub>, and C<sub>max</sub>. If the dose is adjusted in Part 2 of the study the F<sub>rel</sub> calculations will be dose adjusted.
- PK parameters for the hard tablet (fasted) and the dispersible granule formulations (fasted and fed); C<sub>max</sub>, AUC<sub>0-24h</sub>, AUC<sub>0-72h</sub>, AUC<sub>0-168h</sub>, AUC<sub>0-168h</sub>, AUC<sub>0-∞</sub>, time to maximum plasma concentration (T<sub>max</sub>), terminal elimination rate constant (λz), terminal elimination half-life (t<sub>1/2</sub>), apparent volume of distribution during the terminal phase (Vz/F), apparent total plasma clearance (Cl/F), and percentage of AUC that is due to extrapolation from t<sub>last</sub> to infinity (%AUC<sub>extrap</sub>).

# 4 Populations for Analysis

# 4.1 Pharmacokinetic Population

The PK Population will include all subjects who have received at least one dose of IMP and who have a minimum of 1 valid post-dose analytical result for pharmacokinetic parameter estimation. The pharmacokinetic population will be confirmed once all PQP plasma concentration data have been received. The PK population will be used to list and to summarise PK data.

The following PK subsets may also be defined for statistical comparisons;

**PK** subset 1: If any subjects vomit within 4 hours after dosing, their PK data will be assessed, and a decision may be taken to remove these subjects from the statistical comparisons. This would be defined as PK subset 2. This subset will only be deemed necessary if vomiting appears to impact the resulting PK parameters. The generation of this subset will be justified and will be documented formally where needed.

# 5 Pharmacokinetic Data Analysis

# 5.1 Pharmacokinetic Parameter Estimation

The estimation of pharmacokinetic parameters by non-compartmental analysis methods will be performed using Phoenix WinNonlin software (v8.3 or a more recent version, Certara USA, Inc., USA).

# 5.1.1 Imputation of Non-Numerical or Negative Values

The imputation of non-numerical or negative values reported in the input data set will be performed as follows:

- Pre-dose sample times will be entered as zero
- Values that are below the limit of quantification (BLQ) obtained prior to the C<sub>max</sub> will be entered as zero
- Values that are BLQ after the C<sub>max</sub> will be treated as missing
- Values that are quantifiable after at least 2 consecutive BLQ values after C<sub>max</sub> will be treated as missing for the calculation of PK parameters
- Values that are reported as "No Result" or "No Sample" etc. will be treated as missing

# 5.1.2 Rules for Pharmacokinetic Parameter Estimation using WinNonlin

Plasma concentration vs time profiles of PQP (and metabolite) will be generated for each subject. Pharmacokinetic parameters will be estimated using standard Phoenix WinNonlin methods, details of which may be found in the documentation accompanying the WinNonlin software package. The following constraints will apply:

| Parameter Estimation | Constraint |
|---|---|
| Trapezoidal Method | Linear/log trapezoidal rule |
| Number of Points used for Lambda-z | At least 3 post C <sub>max</sub> , not including C <sub>max</sub> |
| Minimum Requirements for AUC | At least 3 consecutive quantifiable concentrations |
| Sampling Times used in analysis | Actual sampling times; when no actual sampling time is available the nominal sampling time will be used |
| Rounded Dose Level | 3 Significant Figures or 2 decimal places |

Where possible, the elimination rate constant (lambda-z) will be calculated for all subjects. The value of lambda-z will be determined by the slope of the regression line of the natural log transformed concentrations vs time.

The choice of data points for determination of lambda-z will be applied by the Phoenix software as a default method, the pharmacokineticist who may adjust the selection in order to provide a more appropriate fit and records of this will be documented in the software data.

# 5.1.3 Data Quality

The following flags/footnotes may be applied to the pharmacokinetic parameters:

| Flag | Footnote |
|---|---|
| a | Rsq of regression was <0.8 |
| b | Extrapolated portion of AUC <sub>(0-inf)</sub> >20% |
| c | Insufficient post-C <sub>max</sub> data points for estimation of lambda-z |
| d | Entire profile BLQ, no pharmacokinetic parameters could be calculated |

In the event that a reliable lambda-z cannot be determined, or the extrapolated portion of  $AUC_{(0-inf)}$  is >20%, then the parameter estimates derived using lambda-z and/or  $AUC_{(0-inf)}$  may be deemed unreliable and excluded from the summary statistics. Additional flags may be applied based on emerging data.

## **5.1.4** Definition of Pharmacokinetic Parameters

The following pharmacokinetic parameters for PQP (and metabolite) in plasma will be estimated where possible and appropriate for each subject and treatment.

**Table 1** Pharmacokinetic Parameters and Reporting Specifications

| Data transfer<br>Term | Parameter | Definition | DP or<br>SF | No. of<br>DP/SF |
|---|---|---|---|---|
| TMAX | $T_{\text{max}}$ | Time at which the maximum observed plasma concentration occurs | DP | 2 |
| CMAX | $C_{\text{max}}$ | Maximum observed plasma concentration | SF | 3 |
| AUC024 | AUC <sub>(0-24)</sub> | Area under the curve from time zero to 24 h | SF | 3 |
| AUC072 | AUC <sub>(0-72)</sub> | Area under the curve from time zero to 72 h | SF | 3 |
| AUC0168 | AUC <sub>(0-168)</sub> | Area under the plasma concentration curve from time zero to 168 hours | SF | 3 |
| AUCLST | AUC <sub>(0-t)</sub> | Area under the plasma concentration curve from time zero up to the last quantifiable concentration | SF | 3 |
| AUCIFO | AUC <sub>(0-inf)</sub> | Area under the curve from time zero extrapolated to infinite time | SF | 3 |
| AUCPEO | %AUC <sub>extrap</sub> | Percentage of AUC that is due to extrapolation from tlast to infinity | DP | 2 |
| LAMZHL | $t_{1/2}$ | Apparent terminal elimination half-life | DP | 2 |
| LAMZ | Lambda-z | Terminal Rate constant | DP | 4 |
| CLFO | CL/F | Apparent total plasma clearance after extravascular administration | SF | 3 |
| VZFO | $V_z/F$ | Apparent volume of distribution during the terminal phase after extravascular administration | SF | 3 |
| FRELCMAX* | Frel C <sub>max</sub> | Relative bioavailability calculated as the ratio of the $C_{max}$ test/ $C_{max}$ reference | DP | 3 |
| FRELAUC72* | Frel AUC <sub>(0-72)</sub> | Relative bioavailability calculated as the ratio of the AUC <sub>(0-72)</sub> test/<br>AUC <sub>(0-72)</sub> reference | DP | 3 |
| FRELAUC168* | Frel AUC <sub>(0-168)</sub> | Relative bioavailability calculated as the ratio of the AUC <sub>(0-168)</sub> test/ AUC <sub>(0-168)</sub> reference | DP | 3 |
| FRELAUCLST* | Frel AUC <sub>(0-t)</sub> | Relative bioavailability calculated as the ratio of the AUC <sub>(0-t)</sub> test/ AUC <sub>(0-t)</sub> reference | DP | 3 |
| FRELAUCINF* DP=decimal places | Frel AUC <sub>(0-inf)</sub> | Relative bioavailability calculated as the ratio of the AUC <sub>(0-inf)</sub> test/ AUC <sub>(0-inf)</sub> reference | DP | 3 |

DP=decimal places SF=significant figures

<sup>\*</sup> The Frel Values will be generated for the comparisons listed in section 4.2. For Part 2 of the study, the calculations may be done on dose corrected parameters if the dose is adjusted in this part of the study.

# 5.2 Statistical Analysis

The relative bioavailability will be assessed for PQP using the ratio of the geometric means for  $AUC_{(0-72)}$ ,  $AUC_{(0-168)}$ ,  $AUC_{(0-inf)}$ , and  $C_{max}$  as follows:

- For Part 1 the comparisons will be Group 2 PQP dispersible granule (320 mg, fasted) [test] over the Group 1 PQP hard tablet (320 mg, fasted) [reference].
- For Part 2 the data from Part 1 Group 2 PQP dispersible granule (320 mg, fasted) will be used as the reference against the following fed test conditions (and dose adjusted where relevant):
  - High-fat meal (Group 3)
  - Low-fat meal representative of African diet (Group 4)
  - Whole milk (Group 5)

A linear mixed effect model will be used to obtain the geometric means ratios, with the logarithm of the PK parameter as response variable, the sequence, treatment and the period as fixed effects, and the subject within sequence as random effect. Least square mean differences (test – reference) will be extracted from the model with two-sided 90% confidence intervals. Mean ratios will be reported with 90% confidence limits after back transformation from the log-scale. The assumption of normality of the distributions will be made when running exploratory bioequivalence analysis.

Bioequivalence analysis will be performed using the Bioequivalence module contained within Phoenix WinNonlin. The following will be selected when analysing the study data

In the Bioequivalence Model tab the following will be selected

- Type of study will be assigned as a Parallel Study
- Type of bioequivalence will be set to Average
- The reference formulation will be set depending on the study part as described above

In the Bioequivalence Fixed effects tab the following will be selected

- Sequence, Formulation and Period are added to the Model specification
- Ln(x) is added to the dependent variables

Normally the random effects are populated however the following should be carried through to this menu

• Subject (Sequence) should be in the random effects model field

Bioequivalence is demonstrated when the 90% confidence interval for parameter is contained between 80 and 125.

# 5.3 Interim Analysis

There will be one interim analysis after dosing of Groups 1 and 2, to review safety data obtained up to Day 15 and PK data obtained up to Day 8, to aid the transition from Part 1 of the study into Part 2.

- For interim analysis purposes the bioanalytical data and generated pharmacokinetic parameters will be tabulated and summarised according to the nominal timepoint in an interim report.
- The following PK parameters for the hard tablet (fasted) and the dispersible granule formulations (fasted) will be generated; C<sub>max</sub>, AUC<sub>0-24h</sub>, AUC<sub>0-72h</sub>, AUC<sub>0-t</sub>, time to maximum plasma concentration (T<sub>max</sub>).
- Interim analysis will be conducted using QC'd data available at the time of analysis and will use nominal sampling timepoints.

Summary statistics (i.e., mean, median, SD, CV%, minimum, maximum, n, geometric mean, geometric SD and geometric CV%) will be calculated for blood concentrations for each time point and treatment. The same will be done for the PK parameters (except  $t_{max}$ ) which will be listed for each individual and summarised by treatment. The  $t_{max}$  summary statistics will be provided as n, minimum, median and maximum only.

Arithmetical mean blood concentration vs. time curve will be produced by treatment on both linear/linear and log10/linear scales. An arithmetic mean comparison plot of tablet fed and granule fed data will also be presented on both linear/linear and log10/linear scales.

Spaghetti plots of individual blood concentrations against nominal sampling times after dosing for each treatment will be produced on both a linear/linear and log10/linear scale. Each subject's concentration profile will be represented on these plots with a different symbol and a legend will be included on the plots to define the symbols used.

Bioequivalence on Part 1 data will be performed as described in section 4.2 for  $C_{max}$ ,  $AUC_{0-72}$  and  $AUC_{0-72}$  and tabulated to form part of the interim PK report.

The interim report will contain a dose recommendation of PQP dispersible granule for use in Part 2 of the study, based upon ensuring that the  $C_{max}$  of PQP granule formulation administered with a high fat meal, will not be predicted to exceed the geometric mean of  $C_{max}$  98 ng/ml with CV 39% obtained from PQP tablet (960 mg) administered in the fasted state (see study MMV\_P21\_01). An assumption will be made that the exposure of PQP in the dispersible granule formulation administered in the fasted state will increase 3-fold when administered with a high fat meal, in line with the exposure increase seen when film-coated tablets (Eurartesim®) are administered with a high fat/high calorie meal.

# **Certificate Of Completion**

Envelope Id: D1D96CF31A204F2E8EA4F45159BA1508

Subject: Complete with DocuSign: PHK2020-174 MMV\_SMC\_22\_01 Pharmacokinetic Data Analysis Plan Version 2...

Source Envelope:

Document Pages: 9 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Signatures: 3

Initials: 0

Envelope Originator: rachael white westwood house 78 Loughborough Rd Quorn, LE12 8Dx

Status: Completed

rachael@Pharmakinetic.co.uk IP Address: 94.192.198.81

**Record Tracking** 

Status: Original

10/2/2023 10:33:48 AM

Holder: rachael white

rachael@Pharmakinetic.co.uk

**Timestamp** 

Location: DocuSign

**Signer Events** Anne Claire Marrast

marrasta@mmv.org

Security Level: Email, Account Authentication

(Required)

anne Claire Marrast

Sent: 10/2/2023 10:35:48 AM Viewed: 10/3/2023 1:51:44 PM Signed: 10/3/2023 1:52:14 PM

Signature Adoption: Pre-selected Style

Signature ID:

Signature

EE083864-2150-49D7-B3D2-7D3273F6C88A

Using IP Address: 217.193.134.164

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 8/11/2021 9:47:14 AM

ID: bf5536ca-fc02-4cdf-8e26-957e53cbef61

Denis Gossen

gossend-consultants@mmv.org

Security Level: Email, Account Authentication

(Required), Logged in

Denis Gossen

Sent: 10/2/2023 10:35:48 AM

Viewed: 10/2/2023 5:34:34 PM

Signed: 10/2/2023 5:36:00 PM

Signature Adoption: Pre-selected Style

Signature ID:

AC827ABF-3B45-4D26-A93B-7F2C91B125E9

Using IP Address: 94.225.233.138

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 5/5/2023 11:29:54 AM

ID: a41729fe-b2ea-408e-8e96-04fabfb2375b

| Signer Events | Signature | Timestamp |
|---|---|---|
| Rachael White | | Sent: 10/2/2023 10:35:49 AM |
| rachael@pharmakinetic.co.uk | Rachael White | Viewed: 10/2/2023 10:36:41 AM |
| Director | | Signed: 10/2/2023 10:37:05 AM |
| Director | Signature Adoption: Pre-selected Style | |
| Security Level: Email, Account Authentication | Signature ID: | |
| (Required) | 2BDFAD0F-F6B3-4023-A90E-30CE7A0ABDD0 | |
| | Using IP Address: 94.192.198.81 | |
| | With Signing Authentication via DocuSign passwore | d |
| | With Signing Reasons (on each tab): | |
| | I approve this document | |
| Electronic Record and Signature Disclosure: | | |

# Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Noton, Frants | | |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Signature<br>Status | Timestamps |
| , | _ | · |
| Envelope Summary Events Envelope Sent Certified Delivered Signing Complete | Status Hashed/Encrypted Security Checked Security Checked | Timestamps 10/2/2023 10:35:49 AM 10/2/2023 10:36:41 AM 10/2/2023 10:37:05 AM |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, director (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

## How to contact director:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: rachael@Pharmakinetic.co.uk

# To advise director of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at rachael@Pharmakinetic.co.uk and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from director

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to rachael@Pharmakinetic.co.uk and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with director

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to rachael@Pharmakinetic.co.uk and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify director as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by director during the course of your relationship with director.